CLINICAL TRIAL: NCT02114164
Title: A Comparative Study of CO2 Exchange Patterns Between Valve-free Trocar (AirSeal®) Versus Standard Trocar (Endopath®) During Robotic Prostatectomies
Brief Title: Study of Carbon Dioxide Exchange Patterns During Robotic Prostatectomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OhioHealth (Other)
Collaborators: SurgiQuest, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OH1-13-00489
Record Dates: First submitted 2014-01-10; First posted 2014-04-15 (Estimated); Results first posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-10

CONDITIONS: Prostate Cancer; Pneumoperitoneum
Keywords: AirSeal; Trocar; Carbon Dioxide Exchange and Absorption
MeSH Terms: conditions — Prostatic Neoplasms; Pneumoperitoneum

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- AirSeal System (Active Comparator): This group receives the AirSeal System for intraoperative insufflation.
  Interventions: Device: AirSeal System
- Standard Endopath (Active Comparator): This group receives the Standard Endopath Trocar for intraoperative insufflation.
  Interventions: Device: Standard Endopath

INTERVENTIONS:
Device: AirSeal System — To analyze the results of patients randomized to either the AirSeal system or Standard Endopath trocar.
  Other Names: Valve-free Trocar
  Arms: AirSeal System
Device: Standard Endopath — This group receives the Standard Endopath Trocar for intraoperative insufflation.
  Other Names: Endopath Trocar
  Arms: Standard Endopath

SUMMARY:
The AirSeal® System will allow for lower carbon dioxide (CO2) absorption rates than the standard Endopath System.

DETAILED DESCRIPTION:
The primary observation to be made is the level of carbon dioxide in the arterial blood, specifically when the patient is insufflated and deflated during the surgery. As a result of the consistent pressure that the AirSeal® system maintains, carbon dioxide will be absorbed in lower levels when compared to the standard of care systems in which fluctuations in intra-peritoneum pressure are seen.

ELIGIBILITY:
Inclusion Criteria:

* Age>18
* Eligible and elect to undergo robotic prostatectomy surgery @ OhioHealth Dublin Methodist Hospital

Exclusion Criteria:

* Age < 18
* Emergency surgery
* Ascites
* BMI>44 or <18

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2016-08; Primary Completion 2018-05-03 (Actual); Study Completion 2019-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronney Abaza, MD,FACS, Principal Investigator — OhioHealth
Locations (1):
- Dublin Methodist Hospital, Columbus, Ohio, United States

REFERENCES:
- [Derived] Abaza R, Martinez O, Murphy C. Randomized Controlled Comparison of Valveless Trocar (AirSeal) vs Standard Insufflator with Ultralow Pneuomoperitoneum During Robotic Prostatectomy. J Endourol. 2021 Jul;35(7):1020-1024. doi: 10.1089/end.2020.1025. Epub 2021 Jan 21. PMID 33349135

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 9 participants withdrew from the study after providing informed consent but before being randomized to a group and receiving an intervention
Period: Overall Study
Arm/Group | AirSeal System | Standard Endopath
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AirSeal System | Standard Endopath | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (5.6) | 62.0 (6.7) | 61.5 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Females not enrolled, as study is about prostate cancer | NA — Females not enrolled, as study is about prostate cancer | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | 50 | 50 | 100
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian | 50 | 42 | 92
  Race/Ethnicity: African American | 0 | 7 | 7
  Race/Ethnicity: Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Data were not recorded for one patient in the Standard Endopath group.
  kg/m^2
    number analyzed (Participants) | 50 | 49 | 99
    (all) | 29.1 (4.3) | 28.3 (3.3) | 28.7 (3.8)
Preoperative hemoglobin [Mean (Standard Deviation); unit: g/dL] — Population: Data not recorded for one participant in the Standard Endopath group
  g/dL
    number analyzed (Participants) | 50 | 49 | 99
    (all) | 15.1 (1.0) | 14.7 (1.0) | 14.8 (1.0)
Preoperative creatinine [Mean (Standard Deviation); unit: mg/dL] — Population: Data not recorded for one participant in the Standard Endopath group
  mg/dL
    number analyzed (Participants) | 50 | 49 | 99
    (all) | 0.89 (0.1) | 0.96 (0.2) | 0.92 (0.1)

OUTCOME MEASURES:

1. Primary Outcome: Intraoperative Pneumoperitoneal Pressure (mmHg)
Description: Pneumoperitoneal pressure is the pressure exerted by air or gas in the abdominal (peritoneal) cavity. As the amount of air/gas increases, the pressure (mmHg) increases. The highest pressure that occurred during the procedure was compared between groups.
Time Frame: Through end of procedure, an average of 156 minutes
Population: Data were missing for one participant in each group.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AirSeal System | Standard Endopath
Number analyzed (Participants) | 49 | 49
mmHg | 7.9 (2.5) | 9.9 (2.9)
Statistical Analysis 1: Comparison: AirSeal System vs Standard Endopath; Test type: Other; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Intraoperative Arterial Blood Gas Carbon Dioxide (mmHg).
Description: The amount of dissolved carbon dioxide (PaCO2) in arterial blood (mmHg) during the operative procedure
Time Frame: Baseline, 60 minutes, and at end of procedure, an average of 156 minutes
Population: Data were missing for one participant in the Standard Endopath group at all time points. Data were missing for two AirSeal participants at baseline and 60 minutes, and for one AirSeal participant at end of procedure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AirSeal System | Standard Endopath
Number analyzed (Participants) | 50 | 49
mmHg
  Baseline: number analyzed (Participants) | 48 | 49
  Baseline | 39.5 (4.9) | 39.2 (5.3)
  60 minutes: number analyzed (Participants) | 48 | 49
  60 minutes | 41.5 (7.7) | 41.2 (5.2)
  End of procedure: number analyzed (Participants) | 49 | 49
  End of procedure | 45.1 (6.1) | 44.1 (5.5)
Statistical Analysis 1: Comparison: AirSeal System vs Standard Endopath; Test type: Other; p = 0.39, t-test, 2 sided

3. Secondary Outcome: End-tidal Carbon Dioxide Pressure (mmHg)
Description: End-tidal carbon dioxide pressure is the partial pressure of carbon dioxide at the end of exhalation. Normal value is 35-45 mmHg.
Time Frame: Baseline, 60 minutes, and at end of procedure, an average of 156 minutes
Population: Missing data for five, five, and seven AirSeal participants at baseline, 60 minutes, and end of procedure, respectively. Missing data for five, four, and four participants at baseline, 60 minutes, and end of procedure, respectively.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AirSeal System | Standard Endopath
Number analyzed (Participants) | 50 | 49
mmHg
  Baseline: number analyzed (Participants) | 45 | 45
  Baseline | 31.47 (3.9) | 29.96 (3.1)
  60 Minutes: number analyzed (Participants) | 45 | 46
  60 Minutes | 32.80 (3.6) | 30.96 (3.2)
  End of procedure: number analyzed (Participants) | 43 | 46
  End of procedure | 34.77 (8.9) | 34.17 (7.2)
Statistical Analysis 1: Comparison: AirSeal System vs Standard Endopath; Test type: Other; p = 0.13, t-test, 2 sided — Comparison at baseline
Statistical Analysis 2: Comparison: AirSeal System vs Standard Endopath; Test type: Other; p = 0.018, t-test, 2 sided — Comparison at 60 minutes
Statistical Analysis 3: Comparison: AirSeal System vs Standard Endopath; Test type: Other; p = 0.712, t-test, 2 sided — Comparison at end of procedure

4. Secondary Outcome: Carbon Dioxide Elimination (mmHg)
Description: Carbon dioxide elimination was calculated using end-tidal carbon dioxide pressure (EtCO2), tidal volume, respiratory rate, barometric pressure (pB = 760mm Hg), partial pressure of water vapor (PH2O = 13 mm Hg), and patient weight (kg)
Time Frame: Baseline, 60 minutes, and at end of procedure, an average of 156 minutes
Population: Missing data for eight, six, and nine AirSeal participants at baseline, 60 minutes, and end of procedure, respectively. Missing data for eight, seven, and eight Standard Endopath participants at baseline, 60 minutes, and end of procedure, respectively.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AirSeal System | Standard Endopath
Number analyzed (Participants) | 50 | 49
mmHg
  Baseline: number analyzed (Participants) | 42 | 42
  Baseline | 3.15 (0.67) | 3.28 (0.64)
  60 minutes: number analyzed (Participants) | 44 | 43
  60 minutes | 3.24 (0.74) | 3.28 (0.6)
  End of procedure: number analyzed (Participants) | 41 | 42
  End of procedure | 3.04 (1.35) | 3.11 (0.65)
Statistical Analysis 1: Comparison: AirSeal System vs Standard Endopath; Test type: Other; p = 0.42, t-test, 2 sided — Comparison at baseline
Statistical Analysis 2: Comparison: AirSeal System vs Standard Endopath; Test type: Other; p = 0.75, t-test, 2 sided — Comparison at 60 minutes
Statistical Analysis 3: Comparison: AirSeal System vs Standard Endopath; Test type: Other; p = 0.99, t-test, 2 sided — Comparison at end of procedure

5. Secondary Outcome: Intraoperative Arterial Blood Gas Oxygen (mmHg).
Description: The amount of dissolved oxygen (PaO2) in arterial blood (mmHg).
Time Frame: Baseline, 60 minutes, and end of procedure, an average of 156 minutes
Population: Data missing for one Standard Endopath participant at all time points. Data missing for two AirSeal participants at baseline and 60 minutes, and one AirSeal participant at end of procedure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AirSeal System | Standard Endopath
Number analyzed (Participants) | 49 | 49
mmHg
  Baseline: number analyzed (Participants) | 48 | 49
  Baseline | 361.9 (79.3) | 364.3 (81.9)
  60 minutes: number analyzed (Participants) | 48 | 49
  60 minutes | 283.9 (115.4) | 294 (105.0)
  End of procedure | 286.5 (99.1) | 290.2 (99.4)
Statistical Analysis 1: Comparison: AirSeal System vs Standard Endopath; Test type: Other; p = 0.88, t-test, 2 sided — Comparison at baseline
Statistical Analysis 2: Comparison: AirSeal System vs Standard Endopath; Test type: Other; p = 0.65, t-test, 2 sided — Comparison at 60 minutes
Statistical Analysis 3: Comparison: AirSeal System vs Standard Endopath; Test type: Other; p = 0.86, t-test, 2 sided — Comparison at end of procedure

6. Secondary Outcome: Number of Ventilator Interventions
Description: The number of times the anesthesiologist had to adjust ventilator settings
Time Frame: Through end of procedure, an average of 156 minutes
Population: Missing data for two participants in the AirSeal group and one participant in the Standard Endopath group
Measure: Mean (Standard Deviation); unit: Count of interventions
Arm/Group | AirSeal System | Standard Endopath
Number analyzed (Participants) | 48 | 49
Count of interventions | 0.69 (1.1) | 0.66 (0.9)
Statistical Analysis 1: Comparison: AirSeal System vs Standard Endopath; Test type: Other — Number of interventions required by the anesthesiologists were compared between the AirSeal and standard Endopath groups using zero-inflated Poisson regression; p = 0.41, Zero-inflated Poisson regression

7. Secondary Outcome: Procedure Time (Minutes)
Description: The duration of the procedure
Time Frame: Through end of procedure, an average of 156 minutes
Population: Missing data for one participant in the AirSeal group and one participant in the Standard Endopath group
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | AirSeal System | Standard Endopath
Number analyzed (Participants) | 49 | 49
Minutes | 158.6 (22.4) | 153.0 (19.9)
Statistical Analysis 1: Comparison: AirSeal System vs Standard Endopath; Test type: Other; p = 0.09, t-test, 2 sided

8. Secondary Outcome: Smoke Evacuation Quality
Description: Smoke evacuation quality throughout the procedure was assessed by the surgeon as below average, average, or above average
Time Frame: Through end of procedure, an average of 156 minutes
Population: Missing data for one participant in the AirSeal group and two participants in the Standard Endopath group
Measure: Count of Participants; unit: Participants
Arm/Group | AirSeal System | Standard Endopath
Number analyzed (Participants) | 49 | 48
Participants
  Below Average | 4 | 16
  Average | 25 | 18
  Above Average | 20 | 14
Statistical Analysis 1: Comparison: AirSeal System vs Standard Endopath; Test type: Other; p < 0.001, Chi-squared

ADVERSE EVENTS:
Time Frame: Through hospital discharge, an average of 8.4 hours
Description: All patients were assessed through discharge for device malfunction, wound infection, urine output, nausea, and vomiting.
Arm/Group | AirSeal System | Standard Endopath
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 1/50 | 3/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AirSeal System (N=50) | Standard Endopath (N=50)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/64/NCT02114164/Prot_SAP_000.pdf